CLINICAL TRIAL: NCT02823236
Title: Efficacy of Intralesional Triamcinolone and 8% Topical Pirfenidone for Treatment of Keloid Scars: 3-arm Trial
Brief Title: Efficacy of Intralesional Triamcinolone and 8% Topical Pirfenidone for Treatment of Keloid Scars
Acronym: LADISLAO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Dermatológico Dr. Ladislao de la Pascua (Other)
Collaborators: Grupo Medifarma, S. A. de C. V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90/15
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Keloid
Keywords: Keloid; Scar
MeSH Terms: conditions — Keloid; Cicatrix | interventions — pirfenidone; Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intralesional Triamcinolone (Active Comparator): A dosage of 4mg/cm2 of intralesional triamcinolone will be injected in the keloid scar every 4 weeks during 6 months.
  Interventions: Drug: Intralesional Triamcinolone
- Topical Pirfenidone (Experimental): Dosage commensurate with scar surface to be treated. After washing and drying the affected area, a thin layer of 8% pirfenidone will be applied on the scar, three times a day, for 6 months.
  Interventions: Drug: Topical Pirfenidone
- Triamcinolone + Pirfenidone (Experimental): A dosage of 4mg/cm2 of intralesional triamcinolone will be injected in the keloid scar every 4 weeks during 6 months. Simultaneously, a thin layer of 8% pirfenidone will be applied on the scar, three times a day, for 6 months.
  Interventions: Drug: Triamcinolone + Pirfenidone

INTERVENTIONS:
Drug: Topical Pirfenidone — Pirfenidone 8% gel will be applied three times per day during 6 months in the surface of the keloid scar.
  Other Names: KitosCell
  Arms: Topical Pirfenidone
Drug: Triamcinolone + Pirfenidone — Triamcinolone will be injected in the keloid scar 4 mg/cm2 every 4 weeks for 6 months. And pirfenidone 8% gel will be applied three times per day during 6 months in the surface of the keloid scar.
  Other Names: Kenalog + KitosCell
  Arms: Triamcinolone + Pirfenidone
Drug: Intralesional Triamcinolone — Triamcinolone will be injected in the keloid scar 4 mg/cm2 every 4 weeks for 6 months.
  Other Names: Kenalog
  Arms: Intralesional Triamcinolone

SUMMARY:
The aim of the study is to assess the efficacy and safety of the combination of intralesional triamcinolone (at doses of 4mg / cm2 at intervals of 4 weeks) and topical pirfenidone 8% (every 8 hours continuously) compared with their isolated application, in the treatment of keloid scars in adults. The duration of this three-arm clinical trial will be 12 months, a 6-month period for treatment and a follow-up of 6 months to assess recurrences. The estimated number of persons to be recruited and randomized for the study is 102.

DETAILED DESCRIPTION:
Individuals with keloid scars will be randomized to 3 arms of treatment in order to assess the efficacy of combining intralesional triamcinolone and topical pirfenidone compared with the isolated application of these drugs. The interventions will last 6 months but the individuals will be assessed monthly to determine recurrences for 6 more months. The scar size will be measure at weeks 12, 24 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Keloids size equal or major than 1 cm
* Keloids less than 5 years old
* Keloids in trunk

Exclusion Criteria:

* Keloid with a surgical indication
* Hypertrophic scars
* Scars after burn wounds
* Pregnancy
* Lactation
* Use of systemic chemotherapeutics or chronic use of systemic corticosteroids or immunosuppressive medication
* Known hypersensitivity for triamcinolone or pirfenidone
* Severe comorbidity not controlled
* Inflammatory acne
* Diabetes Mellitus
* Hypertension
* Renal, hepatic or respiratory failure
* Topical treatment 4 weeks before recruitment
* Previous treatment with intralesional steroids

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2016-10-24 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Keloid Scar Assessment | 0 and 24 weeks
  Assessment using the Vancouver Scar Scale (VSS)
Change in Keloid Scar Assessment by Patients | 0 and 24 weeks
  Assessment using the Patient and Observer Scar Assessment Scale (POSAS)

SECONDARY OUTCOMES:
Occurrence of adverse effects | Every 4 weeks after the beginning of the intervention up to 52 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Quality of life of the patient | 24 weeks
  Dermatology Life Quality Index
Recurrence defined as an increase size of the keloid scar at week 52 | 52 weeks
  Number of patients with an increase size of the keloid scar compared with the size obtained at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Martha Alejandra Morales-Sánchez, MD, MSc, Principal Investigator — Centro Dermatológico Dr. Ladislao de la Pascua
Locations (1):
- Centro Dermatológico "Dr. Ladislao de la Pascua", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided